CLINICAL TRIAL: NCT06375213
Title: Investigating Neurocognitive Disorders Epidemiology
Acronym: INDE
Status: Recruiting | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Principal Investigator, Poosanu Thanapornsangsuth, Doctor, King Chulalongkorn Memorial Hospital
Other Study IDs: 425/66
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dementia; Cognitive Decline; Alzheimer Disease
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease | interventions — Genes, fms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA) plasma and buffy coat, EDTA whole blood, serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cognitively healthy: This cohort includes participants with or without subjective complaints whose results of cognitive examination are normal. Participants will undergo clinical, epidemiological, and cognitive assessments, as well as biospecimen collection every two years, over an 8-year follow-up period.
  Interventions: Diagnostic Test: Plasma tau phosphorylated at Thr217; Other: Neurocognitive examination
- Mild cognitive impairment: This cohort includes participants whose results of cognitive examination are abnormal but have not met the criteria for dementia. Participants will undergo annual clinical, epidemiological, and cognitive assessments, as well as biospecimen collection, for a duration of six years.
  Interventions: Diagnostic Test: Plasma tau phosphorylated at Thr217; Other: Neurocognitive examination
- Late onset dementia: This cohort includes participants with dementia whose symptoms onset after the age of 65. Participants will undergo annual clinical, epidemiological, and cognitive assessments, as well as biospecimen collection, for a duration of two years.
  Interventions: Diagnostic Test: Plasma tau phosphorylated at Thr217; Other: Neurocognitive examination
- Early onset dementia: This cohort includes participants with dementia whose symptoms onset before the age of 65. Participants will undergo annual clinical, epidemiological, and cognitive assessments, as well as biospecimen collection, for a duration of six years.
  Interventions: Diagnostic Test: Plasma tau phosphorylated at Thr217; Other: Neurocognitive examination

INTERVENTIONS:
Diagnostic Test: Plasma tau phosphorylated at Thr217 — Plasma concentration of tau protein phosphorylated at Thr217 as measured on the Meso Scale Discovery, single molecule array (Simoa) or the in-house mass spectrometry platform.
  Other Names: S-PLEX Human Tau (pT217) Kit; ALZpath pTau-217 CARe Advantage Kit
Other: Neurocognitive examination — Traditional (paper and pencil) neurocognitive/neuropsychiatric examination performed by certified psychologists. This includes: Mini Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Clinical Dementia Rating (CDR), Wechsler Memory Scale - Fourth Edition (WMS-IV), Neuropsychiatric Inventory - Questionnaire (NPI-Q), Thai Geriatric Depression Scale (TGDS), General Anxiety Disorder - 7 (GAD-7), The Barthel activities of daily living (ADL) Index, Chula ADL Index.

SUMMARY:
This is a prospective cohort study with the main purpose of predicting progression neurocognitive disorders in Thai population. The main predictor variables to be evaluated are plasma phosphorylated tau (p-tau) level and cognitive test scores, which will be combined using statistical/computational modeling. Additionally, it seeks to evaluate biomarkers for diagnosing disease pathologies, understand their correlation with clinical outcomes, and explore the socioeconomic impact of neurocognitive disorders. The study invites both participants for biospecimen collection, structured interviews, and cognitive examinations and schedules follow-up visits annually or biennially.

DETAILED DESCRIPTION:
The INDE study is a prospective cohort aimed at investigating the natural history and epidemiology of neurocognitive disorders in Thailand. Its primary objective is to develop a predictive model that combines biomarkers (eg. plasma phosphorylated tau) and cognitive performance to accurately predict cognitive decline. Additional objectives include cross-sectional evaluation of various biomarkers for diagnosing disease pathologies, identifying correlations between biomarkers and clinical outcomes, understanding the impact of receiving a biological diagnosis, describing the epidemiology of neurocognitive disorders including risk factors and social determinants of health (SDH), exploring the socioeconomic consequences of these disorders, and establishing a biorepository for future research. The study invites both healthy volunteers and patients referred from memory clinics to participate in a 4-hour visit during which various research procedures are conducted: collection of biospecimens (blood, saliva, sweat), structured interviews covering symptoms, comorbidities, risk factors, SDH, and quality of life, as well as a comprehensive cognitive examination. Participants are scheduled for annual or biennial follow-up visits based on their cognitive status. For those consenting to specific disclosures, investigators provide some biomarker test results and offer post-test counseling based on available research literature. Depending on current funding, a subset of participants meeting additional criteria may also undergo evaluation using appropriate neuroimaging or cerebrospinal fluid (CSF) biomarkers.

ELIGIBILITY:
1. Cognitively Healthy Individuals

   INCLUSION CRITERIA
   * Demonstrate normal cognitive function within the expected range on objective cognitive tests.
   * Proficient in speaking and understanding Thai without the need for a translator to participate.

   EXCLUSION CRITERIA
   * Significant neurological or uncontrolled psychiatric illness.
   * Significant unstable systemic condition or end-stage organ failure that affects study participation.
2. Mild Cognitive Impairment

   INCLUSION CRITERIA
   * Display impaired/abnormal performance on objective cognitive tests.
   * Does not meet criteria for dementia per NIA-AA (or major neurocognitive disorder per DSM-5).
   * Proficient in speaking and understanding Thai without the need for a translator to participate.

   EXCLUSION CRITERIA
   * Significant neurological or uncontrolled psychiatric illness.
   * Significant unstable systemic condition or end-stage organ failure that affects study participation.
3. Late Onset Dementia

   INCLUSION CRITERIA
   * Display impaired/abnormal performance on objective cognitive tests.
   * Meets criteria for dementia per NIA-AA (or major neurocognitive disorder per DSM-5), including dementia due to Alzheimer's disease or other causes.
   * Begins to experience symptoms, identified by the physician as a part of dementia continuum, occurring after the age of 65.
   * Proficient in speaking and understanding Thai without the need for a translator to participate.

   EXCLUSION CRITERIA
   * Significant neurological or uncontrolled psychiatric illness.
   * Significant unstable systemic condition or end-stage organ failure that affects study participation.
4. Early Onset Dementia

INCLUSION CRITERIA

* Display impaired/abnormal performance on objective cognitive tests.
* Meets criteria for dementia per NIA-AA (or major neurocognitive disorder per DSM-5), including dementia due to Alzheimer's disease or other causes.
* Begins to experience symptoms, identified by the physician as a part of dementia continuum, occurring before the age of 65.
* Proficient in speaking and understanding Thai without the need for a translator to participate.

EXCLUSION CRITERIA

* Significant neurological or uncontrolled psychiatric illness.
* Significant unstable systemic condition or end-stage organ failure that affects study participation.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population of this study comprises individuals with a risk of cognitive decline in Thailand categorized by their cognitive status.
Sampling Method: Probability Sample
Enrollment: 990 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2035-08-24 (Estimated); Study Completion 2035-08-24 (Estimated)

PRIMARY OUTCOMES:
Progression to dementia | At 2, 4, 6 and 8 years
  Fulfilling the criteria for dementia according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) 2018 criteria or major neurocognitive disorder (according to DSM-5) as evaluated by neurologist with special interests in neurocognitive disorders. If such designation is not available, reaching a global CDR score of 1 will be used as a substitute. This outcome only applies to cognitively healthy and mild cognitive impairment cohort.
Changes in Sum of Boxes of the Clinical Dementia Rating Scale | At 2, 4, 6 and 8 years
  Administered by a certified psychologist in accordance with Morris, J.C. (1993).
  Minimum value: 0 Maximum value: 18 Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in the Montreal Cognitive Assessment | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 0 Maximum value: 30 Higher scores mean a better outcome.
Changes in the Montreal Cognitive Assessment - Memory Index Score | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 0 Maximum value: 15 Higher scores mean a better outcome.
Changes in the Mini Mental State Examination | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 0 Maximum value: 30 Higher scores mean a better outcome.
Changes in the Wechsler Memory Scale - Fourth Edition (WMS-IV) Visual Reproduction Scaled Score | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 1 Maximum value: 19 Higher scores mean a better outcome.
Changes in the Wechsler Memory Scale - Fourth Edition (WMS-IV) Logical Memory Scaled Score | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 1 Maximum value: 19 Higher scores mean a better outcome.
Changes in the Wechsler Memory Scale - Fourth Edition (WMS-IV) Verbal Paired Associates Scaled Score | At 2, 4, 6 and 8 years
  Administered by a certified psychologist. Minimum value: 1 Maximum value: 19 Higher scores mean a better outcome.
Biological diagnosis of Alzheimer's disease | within 6 months of baseline measurement
  Receiving the diagnosis of Alzheimer's disease based on the abnormality of any pathology-specific biomarkers that fulfills the current NIA-AA criteria. These biomarkers include, but not limited to, amyloid positron emission tomography (PET) (eg. [18 F]-Florbetaben PET), tau-PET (eg. [18F]PI-2620 PET), or CSF levels of core Alzheimer's disease biomarkers.
Biological staging of Alzheimer's disease | within 6 months of baseline measurement
  Staging of Alzheimer's disease based on the abnormality of pathology-specific biomarkers according to the current NIA-AA criteria.
Quantitative amyloid PET uptake. | within 6 months of baseline measurement
  Amyloid PET uptake tracer uptake quantified in Centiloids.
Quantitative tau PET uptake in various cortical regions. | within 6 months of baseline measurement
  Cortical tau-PET uptake measured using mean standardized uptake value ratios of referenced against inferior cerebellar cortex. The pre-specified regions of interest are analogous with Braak staging (as suggested by Cho, H. (2016).):
  Stage I-II, entorhinal cortex; Stage III, parahippocampal and fusiform cortices, and amygdala; Stage IV, inferior and middle temporal cortices; Stage V, inferior parietal, posterior cingulate, lingual, orbitofrontal, insular, supramarginal, lateral occipital, superior temporal, precuneus, superior parietal, superior, middle, and inferior frontal, and anterior cingulate cortices; Stage VI, medial occipital, precentral, paracentral, and postcentral cortices.
Future diagnosis of Alzheimer's disease dementia. | At 2, 4, 6 and 8 years
  All of the following:
  1. Fulfilling the criteria for dementia (NIA-AA 2018) or major neurocognitive disorder (DSM-5) as evaluated by neurologist with special interests in neurocognitive disorders. If such designation is not available, reaching a global CDR score of 1 will be used as a substitute.
  2. Receiving the diagnosis of Alzheimer's disease based on the abnormality of any pathology-specific biomarkers that fulfills the current NIA-AA criteria. These biomarkers include, but not limited to, amyloid-PET (eg. [18 F]-Florbetaben PET), tau-PET (eg. [18F]PI-2620 PET), or CSF levels of core Alzheimer's disease biomarkers.
  3. Conclusion made by a neurologist with special interests in neurocognitive disorders that dementia is predominately due to Alzheimer's disease.

OTHER OUTCOMES:
Quality of life (WHOQOL-BREF) | within 14 days of baseline measurement
  Quality of life as measured by the Thai version of the WHOQOL-BREF questionnaire. The scales of 0-100 were subclassified for each QOL domain (ie. physical, psychological, social and environmental).
Quality of life (EQ-5D-5L) | within 14 days of baseline measurement
  Quality of life as measured by the Thai version of the EQ-5D-5L questionnaire. The raw scores were transformed to utility scores for Thai population as previously suggested (Pattanaphesaj J., 2018).
Number of modifiable risk factors | Three months after disclosing the biomarker results.
  Count data of 0-12. Number of risk factors of the following 12 modifiable risk factors still present in a participant.
  1. Untreated hearing impairment
  2. High depression screening score
  3. Active smoker
  4. Social isolation
  5. Untreated hypertension
  6. Obesity
  7. Untreated diabetes
  8. Physical inactivity quantified by International physical inactivity questionnaire
  9. Alcohol consumption over 21 units per week
  10. Average sleep duration less than 6 hours per night
  11. Low vegetable intake less than 2 servings per week
  12. High red meat or processed meat intake over 5 serving per week

CONTACTS AND LOCATIONS:
Overall Officials: Thiravat Hemachudha, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho H, Choi JY, Hwang MS, Kim YJ, Lee HM, Lee HS, Lee JH, Ryu YH, Lee MS, Lyoo CH. In vivo cortical spreading pattern of tau and amyloid in the Alzheimer disease spectrum. Ann Neurol. 2016 Aug;80(2):247-58. doi: 10.1002/ana.24711. Epub 2016 Jul 8. PMID 27323247
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] American Psychiatric Association. Neurocognitive disorders. In Diagnostic and statistical manual of mental disorders (5th ed.). 2013.
- [Background] Pattanaphesaj J, Thavorncharoensap M, Ramos-Goni JM, Tongsiri S, Ingsrisawang L, Teerawattananon Y. The EQ-5D-5L Valuation study in Thailand. Expert Rev Pharmacoecon Outcomes Res. 2018 Oct;18(5):551-558. doi: 10.1080/14737167.2018.1494574. Epub 2018 Jul 6. PMID 29958008